CLINICAL TRIAL: NCT05679531
Title: Effects of Menthol Gum Chewıng on Postoperatıve Nausea, Vomiting, and Length Of Hospital Stay in Children Undergoing Appendectomy: A Randomızed Controlled Trıal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruya Naz (Other)
Responsible Party: Sponsor-Investigator, Ruya Naz, Nurse, Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RNaz
Record Dates: First submitted 2022-12-08; First posted 2023-01-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Nausea and Vomiting; Hospitalism in Children
Keywords: child; appendectomy; nausea and vomiting; chewing gum; length of hospitalization
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Children in the control group, who met the research criteria, were not applied any procedure other than clinical routine protocol and nursing care. After being brought to the pediatric surgery service, patients with nausea and vomiting were filled out with a questionnaire. The severity of nausea was evaluated with the BARF Scale during nausea and vomiting and 30, 60 and 120 minutes after nausea and vomiting in patients with nausea and vomiting.
- Chewing gum group (Experimental): Starting from the second hour after the child was brought to the clinic after appendectomy, menthol sugar free gum was given to children with nausea and vomiting outside the clinical routine nursing care, as soon as they could chew gum and follow the instructions, and were asked to chew for an average of 15 minutes. The product of a single brand of gum was used. In the first stage, the patient's nausea was evaluated with the BARF nausea scale before the intervention. After filling out the patient information form, the patients who met the research criteria were chewed gum for an average of 15 minutes. During the intervention (between 5-10 minutes), the patient was re-evaluated for nausea with the BARF nausea scale at 30.,60. and 120 minutes after the intervention. Episodes of vomiting were recorded in patients with vomiting.After the quantitative stages of the study were completed, the patient's level of relief was evaluated using a verbal descriptive scale.
  Interventions: Other: intervention

INTERVENTIONS:
Other: intervention — After filling out the patient information form, the patients who met the research criteria were chewed gum for an average of 15 minutes.
  Arms: Chewing gum group

SUMMARY:
The study was conducted as an experimental study to determine the effect of menthol chewing gum application on postoperative nausea, vomiting and hospital stay in children with appendectomy. The population of the study consisted of children aged 7-18 who underwent appendectomy in Bursa Yüksek İhtisas Training and Research Hospital Pediatric Surgery clinic between April and June 2022. In the sample of the study, a total of 60 children (menthol gum group- intervention group=30, control=30) who had postoperative nausea-vomiting, accepted to participate in the study and met the sample selection criteria were included. Starting from the second hour after the child was brought to the clinic after appendectomy, the children in the chewing gum group with nausea and vomiting were chewed gum for an average of 15 minutes. The patients in the study group were not intervened except for routine nursing care. During the chewing gum (between 5-10. minutes), up to 30., 60. and 120. Minutes after the chewing gum.The patient was re-evaluated in terms of nausea with the BARF nausea scale. Episodes of vomiting were recorded in patients with vomiting. After the quantitative stages of the study were completed, the patient's level of relief was evaluated using a verbal descriptive scale. Nausea and vomiting were also evaluated before the patient was discharged.

ELIGIBILITY:
Inclusion Criteria:

* Child and parent's willingness to participate in the research
* The child has no intellectual disability or perception problems.
* Patients who underwent general anesthesia
* Patients who do not develop postoperative complications
* Patients in the 7-18 age group
* Patients who can tolerate chewing gum in the postoperative period
* Patients who like to chew gum
* Patients with nausea and vomiting

Exclusion Criteria:

* Patients with a diagnosis of diabetes
* Patients with teeth and jaw problems
* Patients with menthol allergy
* Patients with irritable bowel syndrome
* Patients with a history of reflux
* Patients whose cognitive level is not suitable
* Patients with a nasogastric tube

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Baxter Retching Faces Scale (BARF) | Pre-procedure (< 1 minute)
  The BARF scale was used to assess the severity of nausea. The primary outcome was nausea and vomiting as assessed by the BARF scale, which is used to measure the severity of postoperative nausea in children. The BARF scale consists of six faces and there is a difference of 2 points between each face. The Baxter Retching Faces (BARF) scale is graded from 0 to 10 points. Evaluation: 1 minute before chewing gum.
Baxter Retching Faces Scale (BARF) | During the procedure fifth Minute
  The BARF scale was used to assess the severity of nausea. The primary outcome was nausea and vomiting as assessed by the BARF scale, which is used to measure the severity of postoperative nausea in children. The BARF scale consists of six faces and there is a difference of 2 points between each face. The Baxter Retching Faces (BARF) scale is graded from 0 to 10 points. Evaluation: During chewing gum ( fifth minute)
Baxter Retching Faces Scale (BARF) | after menthol chewing gum 30 minutes
  The BARF scale was used to assess the severity of nausea. The primary outcome was nausea and vomiting as assessed by the BARF scale, which is used to measure the severity of postoperative nausea in children. The BARF scale consists of six faces and there is a difference of 2 points between each face. The Baxter Retching Faces (BARF) scale is graded from 0 to 10 points. Evaluation: 30 minutes after menthol chewing gum
Baxter Retching Faces Scale (BARF) | after menthol chewing gum 60 minutes)
  The BARF scale was used to assess the severity of nausea. The primary outcome was nausea and vomiting as assessed by the BARF scale, which is used to measure the severity of postoperative nausea in children. The BARF scale consists of six faces and there is a difference of 2 points between each face. The Baxter Retching Faces (BARF) scale is graded from 0 to 10 points. Evaluation: 60 minutes after menthol chewing gum
Baxter Retching Faces Scale (BARF) | after menthol chewing gum (120 minutes)
  The BARF scale was used to assess the severity of nausea. The primary outcome was nausea and vomiting as assessed by the BARF scale, which is used to measure the severity of postoperative nausea in children. The BARF scale consists of six faces and there is a difference of 2 points between each face. The Baxter Retching Faces (BARF) scale is graded from 0 to 10 points. Evaluation: 120 minutes after menthol chewing gum

SECONDARY OUTCOMES:
length of hospitalization | Up to 2 week
  The time from the date of hospitalization to the date of discharge was calculated, Up to 2 week

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No